CLINICAL TRIAL: NCT06078631
Title: Influence of Students Behaviors on Thier Performance and Quality of Life on the OSCE
Brief Title: Influence of Students Behaviors on Performance and Quality of Life on the OSCE
Acronym: ECOPERF
Status: Completed | Type: Observational
Sponsor: Claude Bernard University (Other)
Responsible Party: Principal Investigator, Lilot Marc, Director, Doctor, Claude Bernard University
Other Study IDs: ECOPERF1
Record Dates: First submitted 2023-05-27; First posted 2023-10-12 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Objective Structured Clinical Examination; Performance Anxiety
Keywords: stress; physical activity; sedentarity; sleep; quality of life; coping
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The students behave differentially before an exam. This study aims at determining the influence of all these behaviors on the perceived quality of life of students and their performance during their OSCE.

DETAILED DESCRIPTION:
The students behave differentially before an exam. They can be discriminate, on their sleeping, coping, or physical activity behavior. They also show difference in the number of hours they study by weeks or if they use the services offer by their university.

This study aims at determining the influence of all these behaviors on the perceived quality of life of students and their performance during their OSCE (a major exam).

ELIGIBILITY:
Inclusion Criteria:

* all volontary medical students of the third cycle that came for their exam during the sessions of December and May 2023 from the University of Lyon (Medecine ESt)

Exclusion Criteria:

* no exclusion criteria

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Medical students
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-11 (Actual)

PRIMARY OUTCOMES:
PERFORMANCE | obtained 7 days after the OSCE
  Score at the OSCE exam from 0 to 40 points

SECONDARY OUTCOMES:
SF-12 | obtained one hour after the OSCE
  Overall quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Rode, PhD, Study Chair — UCBL1
Locations (1):
- Marc lilot, Lyon, France

IPD SHARING:
Plan to Share IPD: No